CLINICAL TRIAL: NCT06084637
Title: Randomized Control Trial Comparison Between Intra-articular Infiltrations of PRP, MFAT, and PRP-MFAT in the Treatment of Symptomatic Knee Osteoarthritis.
Brief Title: Comparison Between Intra-articular Infiltrations of PRP, MFAT, and PRP-MFAT in the Treatment of Symptomatic Knee Osteoarthritis.
Acronym: MICROPREP3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCAPHM21_0431
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- autologous microfat (MG) (Experimental): Patient will be hospitalized in outpatient surgery. A blood sample will be collected and a lipoaspiration will be performed under local anesthesia during the same operation by the nurses and the surgeon. Then, biological products will be immediately prepared, and a preparation of autologous MG will be injected intra-articularly by th same surgeon.
  Interventions: Biological: Intra-articular injection of autologous microfat
- Platelet-rich plasma (PRP) (Experimental): Patient will be hospitalized in outpatient surgery. A blood sample will be collected and a lipoaspiration will be performed under local anesthesia during the same operation by the nurses and the surgeon. Then, biological products will be immediately prepared, and a preparation of autologous PRP will be injected intra-articularly by th same surgeon.
  Interventions: Biological: Intra-articular injection of autologous platelet-rich plasma
- Microfat autologous-Platelet-rich plasma (MG-PRP) (Experimental): Patient will be hospitalized in outpatient surgery. A blood sample will be collected and a lipoaspiration will be performed for the preparation during the same operation by the nurses and the surgeon. Then, biological products will be immediately prepared, and autologous microfat associated with a preparation of autologous PRP will be injected intra-articularly by th same surgeon.
  Interventions: Biological: Intra-articular injection of autologous microfat and platelet-rich plasma

INTERVENTIONS:
Biological: Intra-articular injection of autologous microfat — A preparation of autologous microfat (5mL) will be injected intra-articularly.
  Arms: autologous microfat (MG)
Biological: Intra-articular injection of autologous platelet-rich plasma — A preparation of autologous platelet-rich plasma (5mL) will be injected intra-articularly.
  Arms: Platelet-rich plasma (PRP)
Biological: Intra-articular injection of autologous microfat and platelet-rich plasma — A preparation of autologous platelet-rich plasma (5mL) and autologous microfat (5mL) will be injected intra-articularly.
  Arms: Microfat autologous-Platelet-rich plasma (MG-PRP)

SUMMARY:
This research protocol evaluate the efficacity of intra-articular injections of autologous microfat associated with a preparation of autologous PRP, in symptomatic, resistant to first-line medical treatment, degenerative or post-traumatic cartilage lesions of the knee.

The primary objective of this study is to show the superiority of intra-articular injection of autologous microfat combined with autologous PRP preparation compared to injection of microfat or PRP used alone, on the KOOS score at 6 months.

DETAILED DESCRIPTION:
Osteoarthritis is the most widespread joint disease in the world, and one of the most frequent causes of pain and functional disability in Western countries. The incidence of cartilage lesions is constantly on the rise, due to the ageing of the population and the traumas associated with the development of sporting activities.

Recently, the emergence of biotherapies in orthopaedics has led to the development of intra-articular injections of autologous platelet-rich plasma (PRP). Their use has been widespread since 2010, based on the demonstration that platelet-enriched plasma, a concentrate of growth factors, can stimulate cartilage regeneration in vitro and in vivo in preclinical models (Saito, Schmidt, Qi, Tchetina). In addition, PRP administration methods can be optimized: since it is a liquid preparation (platelet suspension), administering it within an interface tissue limits its diffusion and potentiates its trophic effect on the injured cartilage site. Adipose tissue represents the most relevant tissue of interest, as it is a stem cell-rich support tissue with full therapeutic potential, and is easily accessible. Thus, a sample of autologous "microfat" (adipose tissue containing small fat lobules and stem cells, harvested under local anaesthetic by manual liposuction using specific fine sampling cannulas) co-administered at the level of the synovial capsule, could play the role of fluid trophic matrix to the PRP.

The hypothesis of this project is that the standardized injection of an innovative treatment (microgrease and autologous PRP dose) can defer the need for knee arthroplasty in patients with gonarthrosis resistant to first-line medical treatment. The investigators propose to carry out a clinical study in patients with chondral knee lesions resistant to first-line medical treatment, evaluating the benefit during follow-up of treatment with intra-articular injections of microfat and a standardized preparation of autologous PRP or the combination of the 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender, between 20 and 75 year-old.
* Symptomatics degenerativ or post traumatic chondropathy, on at least one of the 3 knee compartments ICRS grade 2, 3 or 4 with VAS>4 and failure of well-conducted medical treatment for at least 1 year (palliative analgesics adapted to the pain, AINS, rehabilitation by a physiotherapist, injections intra-articulaires de corticoïdes et/ou d'acide hyaluronique)
* Varus or valgus less than or equal to 5°.
* BMI greater than 20 (in order to have sufficient fatty tissue)
* Informed consent signed by the patient
* HB > 10g/dl
* Negative beta-HCG at inclusion and effective contraception for patients of childbearing age, for 1 month.
* Beneficiaries of or affiliated to a social security system

Exclusion Criteria:

* Contraindications to MRI : ocular foreign bodies, pacemaker, neurostimulator, cochlear implant, vascular clips, metallic heart valve
* Body mass index (BMI) of less than 20 kg/m2 not allowig to obtain a sufficient quantity of adipose tissue.
* Thrombocytopenia < 150 G/L
* Thrombocytosis > 450 G/L
* Known thrombopathy
* TP=> PR < 70%.
* TCA=> APR > 1.20s
* Anemia HB < 10g/dl
* Positive markers for the following active infectious diseases: HIV 1 and HIV 2 human immunodeficiency virus infection; HTLV I and II virus infection; Hepatitis B virus infection; Hepatitis C virus infection; Syphilis causative agent infection.
* Use of antiplatelet agents, aspirin, anti-vitamin K drugs for less than 15 days.
* Chronic treatment with oral corticosteroids or the use of such treatment less than 2 weeks prior to inclusion
* Intra-articular corticosteroid injection less than 2 months prior to inclusion
* Intra-articular injection of hyaluronic acid less than 2 months prior to inclusion
* Non-steroidal anti-inflammatory drugs less than 15 days prior to inclusion
* Recent fever or infection (bacterial or viral) less than one month old
* Autoimmune diseases
* Inflammatory arthritis
* Immune deficiency
* Ongoing or chronic infectious diseases (viral or bacterial)
* T Malignant tumours or history of malignant tumours less than 5 years prior to inclusion
* Pregnant or lactating women
* Adults protected by law (guardianship or curatorship)
* Patient participating simultaneously in another research project involving the human person
* Minors
* Persons residing in a health or social institution
* Persons in emergency situations
* Persons deprived of liberty
* Persons not covered by the French social security scheme
* Contraindication to local anesthesia and/or surgery
* Allergy to local anesthetics
* Inmates

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
KOOS score at 6 months | 6 months
  KOOS assesses the short- and long-term consequences of knee injuries, as well as the consequences of primary osteoarthritis. It is percentage from 0 to 100. 0 represents extreme problems and 100 represents no problem.

SECONDARY OUTCOMES:
Pain at 1 month | 1 month
  Pain will assassed by a visual anatomy scale from 0 (no pain) to 10 (pain as bad as it could possibly be)
Pain at 3 months | 3 months
  Pain will assassed by a visual anatomy scale from 0 (no pain) to 10 (pain as bad as it could possibly be)
Pain at 12 months | 12 months
  Pain will assassed by a visual anatomy scale from 0 (no pain) to 10 (pain as bad as it could possibly be)
KOOS score at 1 month | 1 month
  KOOS assesses the short- and long-term consequences of knee injuries, as well as the consequences of primary osteoarthritis. It is percentage from 0 to 100. 0 represents extreme problems and 100 represents no problem.
KOOS score at 3 months | 3 months
  KOOS assesses the short- and long-term consequences of knee injuries, as well as the consequences of primary osteoarthritis. It is percentage from 0 to 100. 0 represents extreme problems and 100 represents no problem.
KOOS score at 12 months | 12 months
  KOOS assesses the short- and long-term consequences of knee injuries, as well as the consequences of primary osteoarthritis. It is percentage from 0 to 100. 0 represents extreme problems and 100 represents no problem.
Proportion of treatment failures | 12 months
  Patients are defined as treatment failures if, during the follow-up period, they undergo one of the following procedures on the treated knee, in the absence of intercurrent events: new injection (whatever the product injected), arthroscopy, arthroplasty, etc.
Proportion of arthroplasties not performed in arthroplasty candidates | 12 months